CLINICAL TRIAL: NCT01862302
Title: Haloperidol Prophylaxis in Cardiac Surgery for Patients at Risk for Delirium: A Randomized Placebo-Controlled Pilot Study
Brief Title: Haloperidol Prophylaxis in Cardiac Surgery for Patients at Risk for Delirium
Acronym: HALPCARD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Andre Lamy, Dr Andre Lamy, MD, FRCSC, MHSc, Cardiac Surgeon, McMaster University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HALPCARD-2013
Record Dates: First submitted 2013-05-09; First posted 2013-05-24 (Estimated); Last update posted 2016-09-16 (Estimated); Status verified 2016-09

CONDITIONS: Postoperative Confusion
Keywords: Prevention delirium; Cardiac surgery
MeSH Terms: interventions — Haloperidol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Haloperidol (Active Comparator): Haloperidol 1mg the night before and 1mg the morning of surgery; OR Haloperidol 2mg the morning of surgery
  Interventions: Drug: Haloperidol
- Placebo (Placebo Comparator): 1 dose the night before and 1 dose the morning of surgery; OR 2 doses the morning of surgery
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Haloperidol — 1mg the night before and 1mg the morning of surgery; OR Haloperidol 2mg the morning of surgery
  Other Names: Haldol
  Arms: Haloperidol
Drug: Placebo — 1 dose the night before and 1 dose the morning of surgery; OR 2 doses the morning of surgery
  Arms: Placebo

SUMMARY:
Will the use of prophylactic Haloperidol for patients undergoing open heart surgery reduce the incidence, duration, and severity of post cardiotomy delirium?

DETAILED DESCRIPTION:
Pilot study for feasibility and safety, n = 40, haloperidol 1mg vs. placebo BID administered night before and day of surgery, then continued for total 72hrs post-op, if delirium occurs study drug is stopped and usual standard of care implemented by MRP.

ELIGIBILITY:
Inclusion Criteria:

* Greater than or equal to 70 years of age, undergoing a median sternotomy OR 60-69yrs of age with one or more of the risk factors:

  * TIA/Stroke;
  * Euroscore greater than or equal to 5;
  * abnormal clock draw.

Exclusion Criteria:

* Parkinsonism,
* on any antipsychotic medications pre-op,
* active delirium,
* emergent surgery,
* Haloperidol allergy,
* schizophrenia,
* prolonged QTc.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2013-08; Primary Completion 2015-09 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Feasibility of conducting a trial utilizing low dose Haloperidol use in patients post cardiac surgery | Participants will be followed for the duration of their hospital stay to a maximum of 30 days.
  If a participant does not develop delirium post operatively, then the confusion assessment method (CAM)will be monitored for 24 hours after the study medication ends. Patients will be followed up until seven days or until discharge if no delirium occurs, or if delirium is detected, up to 30 days or until discharge
Safety monitoring of low dose Haloperidol use in patients post cardiac surgery | Participants will be followed for the duration of their hospital stay to a maximum of 30 days
  If a participant does not develop delirium post operatively, then the confusion assessment method (CAM)will be monitored for 24 hours after the study medication ends. Patients will be followed up until seven days or until discharge if no delirium occurs, or if delirium is detected, up to 30 days or until discharge

SECONDARY OUTCOMES:
The incidence of delirium | Participants will be followed for the duration of their hospital stay to a maximum of 30 days
Delirium severity | Participants will be followed for the duration of their hospital stay to a maximum of 30 days
Total length of stay (LOS), with breakdown for intensive care unit (ICU) days and ward days | Participants will be followed for the duration of their hospital stay to a maximum of 30 days
Duration of delirium | Participants will be followed for the duration of their hospital stay to a maximum of 30 days

OTHER OUTCOMES:
An economic analysis will be completed to determine if Haloperidol prophylaxis resulted in any cost savings | Participants will be followed for the duration of their hospital stay to a maximum of 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Andre Lamy, MD, Principal Investigator — McMaster University
Locations (1):
- Hamilton General Site, Hamilton, Ontario, Canada